CLINICAL TRIAL: NCT06569238
Title: The Role of the Microbiome in Diabetic Foot Ulcers
Brief Title: Diabetic Foot Ulcer (DFU) Rapid Pathogen Identification
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Brian Schmidt, Associate Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HUM00251960; K23DK131261 (NIH)
Record Dates: First submitted 2024-08-21; First posted 2024-08-26 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Foot Ulcer; Diabetes Mellitus; Wound
Keywords: Wound Infection; Wound assessments; Wound's microbiome; Next generation sequencing
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Wounds and Injuries; Wound Infection

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to the control and intervention arms using block randomization. Only tissue review will be randomized.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Conventional bacterial culture (Active Comparator): Wound tissue removed will be sent for standard of care evaluation.
  Interventions: Diagnostic Test: Conventional bacterial culture
- Conventional bacterial culture plus rapid diagnostic group (Experimental): Wound tissue removed will be sent for standard of care evaluation as well as rapid diagnostic with metagenomics next generation sequencing (mNGS).
  Interventions: Diagnostic Test: Conventional bacterial culture; Device: Rapid diagnostic group using mNGS technology

INTERVENTIONS:
Diagnostic Test: Conventional bacterial culture — Participants will have DFU ulcer tissue collected and sent to the laboratory (per usual care practices) that includes the use of conventional bacterial culture analysis (i.e., plates).
Device: Rapid diagnostic group using mNGS technology — Participants will have DFU ulcer tissue collected and have metagenomics sequencing performed. The name of the devices listed for this study are the Illumina MiSeq System with MiSeq Reagent Kit V2 from Illumina and the MinION sequencer (Oxford Nanopore Technologies).
  Arms: Conventional bacterial culture plus rapid diagnostic group

SUMMARY:
The purpose of this study is to evaluate the role of rapid diagnosis of pathogens in treatment of infection and wound healing in diabetic foot ulcers. This research is studying the use of a new device of people to learn if metagenomic next generation sequencing (mNGS) techniques technology is a feasible tool that can be used to direct targeted antibiotic therapy in infected diabetic foot ulcers.

Participant's tissue will be randomized to usual care tissue collection and cultures (standard of care) or usual care tissue collection and cultures (standard of care) plus metagenomics next generation sequencing (mNGS). The participant's will not be randomized to any treatment (i.e. antibiotic therapy).

DETAILED DESCRIPTION:
Participants will have tissue taken per standard of care at the baseline visit. In addition, participants will complete of a comprehensive medical history questionnaire, Michigan Neuropathy questionnaires, and have assessments of the foot ulcer or wound. The study team will follow participants for approximately 12 weeks.

Initial antibiotic therapy to treat diabetic foot ulcer infections are determined by participants treating provider and are based on clinical characteristics, drug allergies or sensitivities, and suspected causative pathogen (i.e., bacteria). In this study, the identification of pathogens using mNGS will be given to the treating physician and may result in additional or different antibiotics.

The decision for antibiotic prescription(s) to treat the diabetic foot ulcer infection will be made by treating providers. The antibiotic plan will be updated according to final culture results (usually 4-6 days following culture of tissue). For those participants randomized to the mNGS cohort, the results (usually 24-36 hours following culture of tissue) will be shared with the treating physician. The treating physician may provide additional or different treatment than initially prescribed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes mellitus
* Have an infected DFU with a surface area ≥0.5 square centimeter (cm2)

  o DFU Infection status will be clinically recorded at time of enrollment according to Infectious Disease Society of America (IDSA): mild, moderate, or severe infection
* Have a hemoglobin A1c[HbA1c] of 12% or less as measured within the last 6 months,
* Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

* Pregnant or lactating
* Uncontrolled blood glucose as demonstrated by a HbA1c of greater than 12%
* Bilateral wound or ulcer
* Current infection of Coronavirus disease 2019 (COVID19)
* Unable to provide informed consent or are unwilling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
The percent change in foot ulcer surface area square centimeter (cm2) after 12 weeks of observation for infected diabetic foot ulcers | Baseline, 12 weeks

SECONDARY OUTCOMES:
Percent of clinical resolved infected DFU for infected DFU participants with clinically resolved infection defined as improvement of greater or equal to two clinical signs of infection | Baseline up to 12 weeks
  Clinical signs of infection includes: local swelling or induration, erythema, local tenderness or pain, local warmth, purulent discharge) with no requirement for additional antibiotics upon follow-up appointments.
Total days of antibiotic therapy for the infected DFU participants | Baseline up to 12 weeks
Number of days to infection resolution for the infected DFU participants | Baseline up to 12 weeks
The percentage of participants with an infected DFU at baseline that resolve clinical infection by study week 4 | Baseline to 4 weeks
The percentage of participants with an infected DFU at baseline that undergo a non-traumatic lower extremity amputation during the study. | Baseline up to 12 weeks
The percentage of participants with an infected DFU at baseline that are hospitalized for infection during the study. | Baseline up to 12 weeks
Post study percentage change of wound surface area (cm2). | Baseline up to 12 weeks
Proportion of participants that reach a 50% reduction in surface area (cm2) of the infected DFU | Baseline up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Brian Schmidt, DPM, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No